CLINICAL TRIAL: NCT01878500
Title: Navigation of the Pelvic Floor in Bladder Exstrophy Using Pre-operative MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00069579
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Bladder Exstrophy
Keywords: Bladder exstrophy epispadias complex; Pelvic floor musculature; Intraoperative stereotactic imaging
MeSH Terms: conditions — Bladder Exstrophy; Bladder Exstrophy and Epispadias Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative stereotactic imaging (Experimental): Surgeon will use intraoperative stereotactic imaging with VectorVision® Cranial Guided Image System by Brainlab Inc. to assist in bladder exstrophy closure.
  Interventions: Device: Intraoperative stereotactic imaging with VectorVision

INTERVENTIONS:
Device: Intraoperative stereotactic imaging with VectorVision — Surgeon will use intraoperative stereotactic imaging with VectorVision® Cranial Guided Image System by Brainlab Inc. to assist in bladder exstrophy closure. Prior to the operation a team consisting of pediatric urologist, pediatric radiologists, and a VectorVision rep will use pre-operative MRI to map out specific bony and muscular structures of the pelvic floor. Doing so will allow the pediatric urologist to use these markers intraoperatively to help guide his closure and also allow for future surgeons who use this technology to understand the correct planes to develop for the same surgery.
  Other Names: VectorVision® Cranial Guided Image System by Brainlab Inc.

SUMMARY:
The aim of this study is to investigate the use of intraoperative stereotactic imaging of the pelvic floor musculature during closure of bladder exstrophy.

DETAILED DESCRIPTION:
Much of the long-term success of classic bladder exstrophy closures depends on the initial closure. Several studies have demonstrated that a key to successful initial closure involves deep dissection of the pelvic floor so that the bladder can be placed in the most posterior and inferior position possible. Oftentimes, the need for repeat closure of the abdomen is required if the initial surgeon failed to properly dissect deep enough into the child's pelvic floor. Many surgeons are unfamiliar with the complex anatomy and are unable to verify that they have properly reached the true pelvic floor during this initial surgery. This often leads to failed closures, which result in poor continence rates later in life.

The investigators are attempting to determine the safety and efficacy of the use the Brainlab, Inc. VisionVector® Cranial Image Guided Surgery System during closure of bladder exstrophy. The value of this research is two-fold. Firstly, the project will help us to verify if the investigators are indeed dissecting down to the proper plane required for successful initial closure of bladder exstrophy. Secondly, this project will help others with relatively less experience with bladder exstrophy to properly identify where they are anatomically during closure of exstrophy, thus yielding higher success rates and better patient care at other centers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-7 years
2. Diagnosis of classic bladder exstrophy
3. Scheduled to undergo bladder exstrophy closure by the principal investigator at Johns Hopkins Hospital's Broadway campus.
4. All eligible participants will be children whose parents or legally authorized representatives have already agreed and are being scheduled for osteotomy and bladder exstrophy closure as determined by their pediatric urologist.
5. Parent or legally authorized representative who is, in the opinion of the investigator, reliable and willing to make themselves and patient available for the duration of the study.
6. Parent or legally authorized representative is able to complete and sign the informed consent document.
7. Patient judged by the investigator to have bladders of sufficient size and elasticity to be suitable for immediate closure as evidenced by the PI's assessment of the patient's bladder template [16].
8. Patient with cardiopulmonary function sufficient to tolerate general anesthesia as evidenced by the pediatrician's and anesthesiologists assessment of the patient's overall cardio-pulmonary status.
9. Patients requiring ferromagnetic metal objects such as a metal pace maker during the OR procedure.

Exclusion Criteria:

1. Lack or withdrawal of consent for primary operative procedure.
2. Parent or legally authorized representative who is, in the opinion of the investigator, not reliable or unwilling to make themselves and patient available for the duration of the study.
3. Parent or legally authorized representative who is unable to understand, complete and/or sign the informed consent document. Non-English speaking parents will automatically be excluded if they are unable to read and understand the consent form.
4. Patient who will not undergo osteotomy prior to closure for any reason

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Gearhart, MD, Principal Investigator — Brady Urological Institute, Department of Pediatric Urology
Locations (1):
- Brady Urological Institute. Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients with bladder exstrophy were recruited. Those who were undergoing exstrophy closure with pelvic osteotomy were included. Those who did not have planned pelvic osteotomy prior to closure were excluded (1).
Period: Overall Study
Arm/Group | Intraoperative Stereotactic Imaging
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Stereotactic Imaging
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] | 28.6 [0.9 to 287.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All patients referred to Johns Hopkins for bladder exstrophy were enrolled at Johns Hopkins in Baltimore, MD.
  Participants
    United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Success or Failure of Exstrophy Closure
Description: A failed bladder closure was defined as bladder prolapse, dehiscence, outlet obstruction, persistent vesicourethral fistula, or a combination of these, or a complication that required repeat closure.
Time Frame: 2 years
Population: 3 patients were simple cystectomies and thus did not represent bladder closures and were subsequently excluded from final analysis.
Measure: Number; unit: exstrophy closures
Arm/Group | Intraoperative Stereotactic Imaging
Number analyzed (Participants) | 44
exstrophy closures
  Successful | 44
  Failed | 0

2. Secondary Outcome: Urinary Continence
Description: Continence rates as determined by total dry time during the day, number of incontinent episodes, and need for dry pads.
Time Frame: 2 years
Population: Data was not collected.
Arm/Group | Intraoperative Stereotactic Imaging
Number analyzed (Participants) | 0

3. Secondary Outcome: Operative Time
Description: Time (measured in minutes) of operation.
Time Frame: Intraoperatively
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intraoperative Stereotactic Imaging
Number analyzed (Participants) | 44
minutes | 619 [503 to 647]

4. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay (in days) for each participant.
Time Frame: Up to 2 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intraoperative Stereotactic Imaging
Number analyzed (Participants) | 44
days | 50 [45 to 54]

5. Secondary Outcome: Peri-operative Complications as Assessed by the Total Number of Transfusions
Description: Peri-operative complications were those encountered immediately before, during, or immediately following the case, primarily regarding need for blood transfusions. Though these are not complications (and deemed necessary/inherent to the operation), they are tracked closely as an outcome measure.
Time Frame: Intraoperatively
Population: as for outcome 1
Measure: Number; unit: transfusions
Arm/Group | Intraoperative Stereotactic Imaging
Number analyzed (Participants) | 44
transfusions | 26

6. Secondary Outcome: Subjective Improved Identification of the Pelvic Floor Anatomy During Bladder Exstrophy Closure as Reported by the Surgeon
Description: Surgeon's were surveyed post-operatively on whether the intervention improved identification of pelvic floor anatomy.
  Measure: Binary, 'Yes' and 'No'
Time Frame: Intraoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Stereotactic Imaging
Number analyzed (Participants) | 44
Participants
  Yes | 44
  No | 0

7. Secondary Outcome: Total Number of Post-operative Complications
Description: Post-operative complications were graded on the Clavien-Dindo Classification System. The Clavien-Dindo System is a standardized classification for reporting and registering complications. It grades the severity of a complication based on the therapy required to treat the complication. It is a tiered system with subdivided categories as follows:
  Grade I and II are considered minor, Grade III is considered moderate and Grades IV and V are severe complications.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: Post-operative complications
Arm/Group | Intraoperative Stereotactic Imaging
Number analyzed (Participants) | 44
Post-operative complications
  Overall complications | 10
  Grade I | 3
  Grade II | 3
  Grade IIIb | 4

ADVERSE EVENTS:
Time Frame: 2 years
Description: Complications were graded on the Clavien-Dindo Classification Scheme to stratify minor from major complications. 3 patients were simple cystectomies and thus did not represent bladder closures and were subsequently excluded from final analysis.
Arm/Group | Intraoperative Stereotactic Imaging
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 10/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraoperative Stereotactic Imaging (N=44)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) — Wound Dehiscence, breakdown
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) — Acute renal injury as determined by rise in Cr, drop-off in urine output
Wound infection (Infections and infestations) | 4 (4) — Infected surgical site
Pin site infection (Infections and infestations) | 1 (1)
Urine leak (Renal and urinary disorders) | 1 (1)
Ureteral obstruction (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT01878500/Prot_SAP_001.pdf